CLINICAL TRIAL: NCT05448768
Title: Biomarker-based Prediction of Cognitive Effects and Potential Mechanisms of Theta-burst Stimulation (TBS) in Subjects With Mild Cognitive Impairment (MCI)
Brief Title: Cognitive Effects and Potential Mechanisms of TBS in Subjects With MCI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202102037A3A0
Record Dates: First submitted 2022-06-27; First posted 2022-07-07 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; theta-burst stimulation; repetitive transcranial magnetic stimulation (rTMS)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The investigators will perform standard intermittent TBS (iTBS) parameters to left DLPFC of every patient in the study. The frequency parameters of TBS are 3-pulse 50-Hz bursts, every 200 ms at 5 Hz, and the intensity is 90% of active motor threshold. A single session of iTBS contains 2 s of TBS repeated every 10 s for 20 times. In this study, we will give two sessions of iTBS separated by 15 min.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amyloid-positive MCI (Active Comparator): The subjects will receive active stimulation of standard intermittent TBS (iTBS) protocol.
  Interventions: Device: TBS for Amyloid-positive MCI
- Amyloid-negative MCI (Active Comparator): The subjects will receive active stimulation of standard intermittent TBS (iTBS) protocol.
  Interventions: Device: TBS for Amyloid-negative MCI

INTERVENTIONS:
Device: TBS for Amyloid-positive MCI — The investigators will perform standard intermittent TBS (iTBS) parameters to left DLPFC of every patient in the study. The frequency parameters of TBS are 3-pulse 50-Hz bursts, every 200 ms at 5 Hz, and the intensity is 90% of active motor threshold. A single session of iTBS contains 2 s of TBS repeated every 10 s for 20 times. In this study, The investigators will give two sessions of iTBS separated by 15 min.
  Arms: Amyloid-positive MCI
Device: TBS for Amyloid-negative MCI — The investigators will perform standard intermittent TBS (iTBS) parameters to left DLPFC of every patient in the study. The frequency parameters of TBS are 3-pulse 50-Hz bursts, every 200 ms at 5 Hz, and the intensity is 90% of active motor threshold. A single session of iTBS contains 2 s of TBS repeated every 10 s for 20 times. In this study, The investigators will give two sessions of iTBS separated by 15 min.
  Arms: Amyloid-negative MCI

SUMMARY:
This study aims to examine the effects and potential mechanisms of theta-burst stimulation (TBS) on cognitive function in individuals with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
The investigators apply the NIA-AA criteria to subtype different endophenotypes of biomarker-defined MCI individuals. This is a prospective, open-label clinical trial, and combined functional neuroimaging study of 18F-FDG-PET to further explore the potential mechanisms. A total of 80 MCI patients will be consecutively recruited and be subjected to iTBS for 5 daily interventions per week for two consecutive weeks. Cognitive evaluation will be performed before and immediately after TBS intervention, and 8 weeks after TBS. Data on functional neuroimaging will be also collected before and after TBS protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 50-90 year
2. Subjects meet Petersen's criteria for mild cognitive impairment (Petersen, Smith et al. 1999)
3. The CDR of MCI patients can be 0-0.5
4. Amyloid PET should ever be performed

Exclusion Criteria:

1. Any subject has a definite diagnosis of epilepsy or history of seizure attack.
2. Current or past history of clinically significant neurological insults affecting brain structure or function like completed stroke, head injury or brain tumor.
3. Any subject has clinically significant or unstable medical diseases including metabolic, renal,liver, lung or cardiovascular disorders including metabolic, renal, liver, lung or cardiovascular disorders.
4. Any subject has current alcohol or other substances abuse and/ or dependence within the recent one year, or prolonged history of major psychiatric disorder like schizophrenia,bipolar disorder, and previously prolonged substances abuse.
5. Any females who is pregnant or lactating.
6. General MRI, TMS and/or PET exclusion criteria including subjects who had received brain aneurysm surgery, or implanted pacemaker, mechanical valves, cochlear implant or other metal devices/ objects that are not MR compatible in the body.

Withdrawal criteria

1. Complications onset after intervention that affect efficacy and safety judgments.
2. New onset or progression of disease that may affect outcomes.
3. Use of other therapies or drugs during the intervention period to change cognitive functions.
4. Any subjects who are recognized as high risk of adverse effects by principle investigator.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination ( MMSE ) | Baseline and immediately after 2 weeks of TBS and 8-week follow-up after TBS
  Change from baseline Mini-Mental State Examination total scores immediately after TBS intervention
Montreal Cognitive Assessment | Baseline and immediately after 2 weeks of TBS and 8-week follow-up after TBS
  Change from baseline Montreal Cognitive Assessment total scores immediately after TBS intervention

SECONDARY OUTCOMES:
The standard uptake values changes of FDG-PET | Before and immediately after TBS intervention
  The standard uptake values (SUV) changes of cerebral glucose metabolism using 18F-FDG-PET

CONTACTS AND LOCATIONS:
Overall Officials: KUAN YI WU, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No